CLINICAL TRIAL: NCT06690593
Title: Gut Microbiota Profiling in Patients With Monoclonal Gammopathy: Implications for Disease Pathogenesis and Progression
Brief Title: Characteristics and Clinical Significance of Gut Microbiota in Patients With Monoclonal Gammopathy
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZhujiangGMMGUS
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-07

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance (MGUS); Intestinal Flora; Multiple Myeloma; M-Protein
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Monoclonal gammopathy patients: (I) Inclusion Criteria:
  1. Age 45 years or older.
  2. Positive screening for monoclonal protein by MALDI-TOF MS.
  3. Meeting the International Classification of Diseases, 11th Revision (ICD-11) criteria for one of the following disease types:Infectious diseases，Tumors，Blood or hematopoietic organ diseases，Immune system diseases，Endocrine, nutritional, or metabolic diseases，Nervous system diseases，Circulatory system diseases，Respiratory system diseases，Digestive system diseases，Musculoskeletal or connective tissue diseases，Urinary and reproductive system diseases.
  4. Sufficient whole blood, plasma, serum, and stool samples available, with relevant case data provided.
  (II) Exclusion Criteria:
  1. History of intestinal tumors, irritable bowel syndrome, or inflammatory bowel disease, or diagnosed during hospitalization.
  2. Antibiotic treatment in the past month.
  3. Insufficient sample volume, or severe hemolysis, lipemia, jaundice, or other unqualified sample conditions.
- Non-monoclonal gammopathy patients: (I) Inclusion Criteria:
  1. Age 45 years or older.
  2. Negative screening for monoclonal protein by MALDI-TOF MS.
  3. Patients meeting ICD-11 criteria for one of the following disease types:Infectious diseases，Tumors，Blood or hematopoietic organ diseases，Immune system diseases，Endocrine, nutritional, or metabolic diseases，Nervous system diseases，Circulatory system diseases，Respiratory system diseases，Digestive system diseases，Musculoskeletal or connective tissue diseases，Urinary and reproductive system diseases.
  4. Sufficient whole blood, plasma, serum, and stool samples available, with relevant case data provided.
  (II) Exclusion Criteria:
  1. History of intestinal tumors, irritable bowel syndrome, or inflammatory bowel disease, or diagnosed during hospitalization.
  2. Antibiotic treatment in the past month.
  3. Insufficient sample volume, or severe hemolysis, lipemia, jaundice, or other unqualified sample conditions.
- Healthy control group: (I) Inclusion Criteria:
  1. Age 45 years or older.
  2. Negative screening for monoclonal protein by MALDI-TOF MS.
  3. No significant diseases found upon medical examination, and confirmed not to have any diseases related to this study.
  4. Sufficient whole blood, plasma, serum, and stool samples available, and relevant case data can be provided.
  (II) Exclusion Criteria:
  1. History of intestinal tumors, irritable bowel syndrome, or inflammatory bowel disease, or diagnosed during hospitalization.
  2. Antibiotic treatment received in the past month. Presence of severe systemic diseases, including malignant tumors.
  3. Insufficient sample volume, or presence of severe hemolysis, lipemia, jaundice, or other unqualified sample conditions.

SUMMARY:
This is an observational case-control study, aiming to systematically analyze the gut microbiome characteristics of patients with monoclonal gammopathy of undetermined significance (MGUS). The study will collect blood and stool samples from MGUS patients, non-MGUS patients (with similar diseases), and healthy controls, and perform multi-omics detection including microbiomics, peptidomics, and biochemical immunology. It will comprehensively analyze the abnormal features of the gut microbiome in MGUS patients, which may help provide new biomarkers and potential mechanisms for the diagnosis, prognosis evaluation, and treatment strategies of MGUS.

DETAILED DESCRIPTION:
This is a case-control, observational single-center study aiming to investigate the impact of common comorbidities on gut microbiome structure and disease progression in patients with monoclonal gammopathy. We plan to collect samples from 11 disease categories, with each category including two groups (monoclonal gammopathy and non-monoclonal gammopathy), as well as 700 age- and gender-matched healthy controls, for a total of 2,990 samples. At enrollment, we will collect whole blood, plasma, serum, and fecal samples from the study participants, and obtain relevant information such as demographic characteristics, lifestyle, family medical history, and medication use.We will perform metagenomic, proteomic, and serum biochemical and immunological analyses on the samples to directly obtain association data between gut microbiome characteristics (as exposure factors) and clinical outcomes (as endpoints). This study will systematically analyze the dysbiosis characteristics of the gut microbiome in monoclonal gammopathy patients, identify key microbial biomarkers, and compare the microbiome structure and clinical laboratory indices between MGUS patients and different comorbidity subgroups, to explore their impact on the disease diagnostic model.

ELIGIBILITY:
(I) Inclusion Criteria:

1. Age 45 years or older;
2. Negative screening for monoclonal protein by MALDI-TOF MS;
3. No significant diseases found upon medical examination, and confirmed not to have any diseases related to this study;
4. Sufficient whole blood, plasma, serum, and stool samples available, and relevant case data can be provided.

(II) Exclusion Criteria:

1. History of intestinal tumors, irritable bowel syndrome, or inflammatory bowel disease, or diagnosed during hospitalization;
2. Antibiotic treatment received in the past month; Presence of severe systemic diseases, including malignant tumors;
3. Insufficient sample volume, or presence of severe hemolysis, lipemia, jaundice, or other unqualified sample conditions.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients aged 45 years and older who meet the following inclusion criteria:
  1. Confirmed negative for monoclonal immunoglobulin by MALDI-TOF MS screening.
  2. No significant diseases found upon medical examination, and confirmed not to have any diseases related to this study.
  3. Availability of sufficient whole blood, plasma, serum, and fecal samples, as well as relevant case information.
  Exclusion criteria include:
  1. History of intestinal tumors, irritable bowel syndrome, or inflammatory bowel disease.
  2. Received antibiotic treatment within the last month.
  3. Presence of severe systemic diseases, including malignant tumors, insufficient sample volume, or presence of sample failure (e.g., severe hemolysis, lipemia, or jaundice).
Sampling Method: Non-Probability Sample
Enrollment: 2990 (Estimated)
Dates: Start 2024-12-26 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
M-protein detection | 24 months
  Plasma samples from all patients will be screened and qualitatively analysed for M proteins using MALDI-TOF MS to determine the presence of patients with monoclonal gammaglobulinemia.
microbiome | 24 months
  To assess the value of the microbiome in predicting the prognosis of patients with monoclonal gammopathy and in diagnosing co-morbidities. To analyse the microbial composition of patient stool samples using 16S rRNA gene sequencing and metagenomics.
metabonomics | 24 months
  To assess changes in plasma metabolomics in patients with monoclonal gammaglobulinaemia. Metabolomics is a large-scale study of small molecules such as fatty acids, bile acids, and lipid mediators.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Professor, Study Chair — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No